CLINICAL TRIAL: NCT00001994
Title: A Pilot Study of 566C80 for the Salvage Treatment of Toxoplasmic Encephalitis in Patients Infected With the Human Immunodeficiency Virus (HIV) Who Have Failed or Are Intolerant of Pyrimethamine-Sulfadiazine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 101A; 02
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1992-03

CONDITIONS: Toxoplasmosis, Cerebral; HIV Infections
Keywords: Toxoplasmosis; AIDS-Related Opportunistic Infections; Naphthoquinones; Encephalitis; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Toxoplasmosis, Cerebral; HIV Infections; Toxoplasmosis; AIDS-Related Opportunistic Infections; Encephalitis; Acquired Immunodeficiency Syndrome | interventions — Atovaquone

INTERVENTIONS:
Drug: Atovaquone

SUMMARY:
To evaluate the safety and tolerance of atovaquone (566C80) in AIDS patients with central nervous system (CNS) toxoplasmosis. To evaluate the efficacy of 566C80 in the acute treatment and suppression of CNS toxoplasmosis in AIDS patients who fail or who cannot tolerate conventional therapy.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following:

* Presumptive diagnosis of AIDS.
* Cerebral toxoplasmosis.
* Expected survival of at least four weeks without therapy.
* Willing and able to give informed consent.

Prior Medication:

Allowed:

* Pyrimethamine-sulfonamide.
* Clindamycin-sulfonamide.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Significant emotional disorder or psychosis.
* Evidence of significant malabsorption, ileus or significant emesis at entry which would inhibit drug absorption.
* Other known central nervous system lesions such as lymphoma, tuberculoma, cryptococcoma, active neurosyphilis. Unwilling or unable to take 566C80 with a meal, enteral supplements (eg:
* Ensure Plus) or pulverized form through a nasogastric tube.
* Active drug or alcohol abuse sufficient in the investigator's opinion to prevent compliance with the study regimen.

Concurrent Medication:

Excluded:

* Drugs with potential anti-toxoplasmosis activity including sulfone, sulfonamide, trimethoprim, pyrimethamine and clindamycin during the acute therapy phase of the trial.
* First three weeks of treatment:
* Retrovir (zidovudine) or any investigational agent including antiretroviral agents (eg:
* ddI,ddC).

Patients with the following are excluded:

* Significant emotional disorder or psychosis.
* Evidence of significant malabsorption, ileus or significant emesis at entry which would inhibit drug absorption.
* Other known central nervous system lesions such as lymphoma, tuberculoma, cryptococcoma, active neurosyphilis. Unwilling or unable to take 566C80 with a meal, enteral supplements (eg:
* Ensure Plus) or pulverized form through a nasogastric tube.
* Active drug or alcohol abuse sufficient in the investigator's opinion to prevent compliance with the study regimen.

Active drug or alcohol abuse sufficient in the investigator's opinion to prevent compliance with the study regimen.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (22):
- United States (18):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Infectious Disease Med Group, Oakland, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF - San Francisco Gen Hosp, San Francisco, California
  - Davies Med Ctr, San Francisco, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Infectious Disease Research Consortium of Georgia, Atlanta, Georgia
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Beth Israel Med Ctr, New York, New York
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - SUNY / Health Sciences Ctr at Stony Brook, Stony Brook, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Gathe, Joseph, M.D., Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Infectious Disease Physicians Inc, Annandale, Virginia
- Canada (4):
  - Southern Alberta HIV Clinic / Foothills Hosp, Calgary, Alberta
  - Dr Julio S G Montaner, Vancouver, British Columbia
  - Wellesley Hosp, Toronto, Ontario
  - Dr Emil Toma / Hotel Dieu de Montreal, Montreal, Quebec

REFERENCES:
- [Background] Masur H, et al. 566C80 is effective as salvage treatment for toxoplasma encephalitis. Int Conf AIDS. 1991 Jun 16-21;7(2):30 (abstract no WB31)